CLINICAL TRIAL: NCT07117110
Title: Plasma Lycopene Concentration as a Dietary Compliance Biomarker - a Pilot Study
Brief Title: Lycopene as a Dietary Compliance Biomarker
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Lionne Venderbos, Assistant Professor, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MEC-2023-0633; NL85468.078.23 (Other: Erasmus MC)
Record Dates: First submitted 2025-07-25; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: lycopene; life style; healthy; male; prostate
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - supplement, tomato soup (Experimental): Group A will take 40 mg lycopene (2,5 pills of food supplement Vitabiotics Ultra Lycopene 15mg, potent extract) first. After a wash-out period, group A will continue and take 250ml of tomato soup (matching with 40mg lycopene) with 20ml olive oil.
  Interventions: Dietary Supplement: Supplement; Other: Tomato soup
- Group B - tomato soup, supplement (Experimental): Group B will take 250 ml of tomato soup (matching with 40 mg lycopene) with 20 ml olive oil first. After a wash-out period, group B will continue and take 40mg lycopene (2,5 pills of food supplement Vitabiotics Ultra Lycopene 15mg, potent extract).
  Interventions: Dietary Supplement: Supplement; Other: Tomato soup

INTERVENTIONS:
Dietary Supplement: Supplement — Group will take 40 mg lycopene (2,5 pills of food supplement Vitabiotics Ultra Lycopene 15mg, potent extract).
Other: Tomato soup — Group will take 250 ml of tomato soup (matching with 40 mg lycopene) with 20 ml olive oil.

SUMMARY:
Rationale: To determine the plasma lycopene concentration before and after an oral intake of lycopene in order to use this measurement as a life style compliance marker.

Objective: Primary objective: to determine if a plasma lycopene concentration can serve as a response parameter after a single dose of dietary lycopene.

Study design: Cross-over interventional pilot study.

Study population: Ten male healthy volunteers 18-75 years. Intervention: Oral food supplement tablet 40 mg lycopene once, versus oral soup of cooked tomatoes equivalent to 40 mg lycopene content. In addition, the participants' habitual diet and actual food intake during the intervention will be measured using a food frequency questionnaire and a food diary.

Main study parameters/endpoints: Variation of plasma lycopene 1 hour before, and 1,3,6,12,24,48,72 hours after intervention.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Eight blood samples of 6 ml full venous blood obtained by vena puncture per intervention per individual, 2 times in a cross-over pilot study, in which interventions are 3 weeks apart (so 2 x 8 samples in 10 volunteers). Risk of vena puncture is negligible, idemque the burden.

ELIGIBILITY:
Inclusion Criteria:

* Male;
* Healthy;
* 18-75 yrs old.

Exclusion Criteria:

* Allergic for tomatoes;
* Any gastrointestinal disorder within 3 months prior to the intervention;
* Recent medication or supplement use;
* Recent substantial change in weight;
* Adherence to a specific diet ( for example the Moorman-diet);
* Using recreational drugs more than once a month;
* Smoking and excessive alcohol consumption (>10 standardized glasses a week).
* Risk of a dependency situation with the researchers.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males by birth.
Enrollment: 10 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To measure lycopene concentration after a single dose of dietary lycopene. | From enrollment until 72 hours after, wash out period of 3 weeks, then again start until 72 hours later.

SECONDARY OUTCOMES:
To measure lycopene concentration after taking a food supplement tablet lycopene of 40mg of lycopene. | Start intervention until 72 hours later, wash-out period, start intervention until 72 hours later.
To measure prior food consumption using a daily food questionnaire. | One week before the dietary intervention a daily food questionnaire will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Lionne DF Venderbos, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT07117110/Prot_000.pdf